CLINICAL TRIAL: NCT03454854
Title: Effectiveness of the Application on Individualized Antithrombotic Therapy in Chinese Patients With Coronary Artery Disease
Brief Title: Effectiveness of the Application(APP) on Individualized Antithrombotic Therapy
Acronym: APP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jiyan Chen, professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDCR2017144H
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Antithrombotic
Keywords: risk evaluation; individualized treatment; coronary artery disease; antithrombotic therapy; Chinese people; Application
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APP-assisted anti-thrombotic therapy (Experimental): Intelligent response system:real-time receiving data or events that doctor or patient terminal upload,then spontaneously evaluate the thrombosis and bleeding risk based on code of point built-in,respectively send messages to doctor and patient after this, then doctors direct the patients to adjust treatment schedule.Develop an exemplary anti-thrombotic therapy network data platform and a intelligent terminal APP, establish an new pattern used in long-time anti-thrombotic management based on dynamic risk evaluation, and promoted and verified by 10 thousands large sample's cohort study.
  Interventions: Device: intelligent terminal APP

INTERVENTIONS:
Device: intelligent terminal APP — Applications(APP) support patients to upload the primary data contain pictures and wearable devices data. When risk-rating changes or serious adverse events(SAE) take place, APP will alert patients to seek medical advice or make a call with the doctor. Beside, terminal of patients furnishes functions like answering frequently asked questions,self-assessment of physical condition,push rehabilitation knowledge etc.

SUMMARY:
Develop an exemplary anti-thrombotic therapy network data platform and a intelligent terminal application(APP), establish an new pattern used in long-time anti-thrombotic management based on dynamic risk evaluation, and promoted and verified by 10 thousands large sample's cohort study.

DETAILED DESCRIPTION:
1.1.Develop and optimize antithrombotic therapy network data platform and thrombotic risk evaluate the intelligent terminal APP, establish a new pattern based on dynamic risk evaluation and event-triggered response, settle the conundrum in clinical practice about antithrombotic therapy such as poor compliance, lag and unreasonable in drug adjustment.

1.2.Settle the technical problem that intelligent terminal APP code isn't compatible with most tablet PCs and smartphones.

1.3.Impel the data platform to render and integrate with the daily medical system, enhance its accuracy, compatibility, privacy, and quality standard.

1.4.Promote the new pattern of anti-thrombotic management by large sample's cohort study, increase the patients' compliance, reduce the readmission rate and adverse event rate of heart and cerebral vessels.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years;
* clinical confirmed coronary heart disease. Including definite history of myocardial infarction, stable angina with exercise electrocardiography test(treadmill exercise) positive, unstable angina with electrocardiogram(ECG) ischemic changes or troponin positive, coronary angiography(CAG) hints at least one coronary artery stenoses over 50%, post-operative of percutaneous coronary intervention(PCI) or coronary artery bypass grafting(CABG);
* Be receiving anti-thrombotic therapy;
* Be voluntary to participate in the study., and sign informed consent form.

Exclusion Criteria:

* inability to obtain consent from participants;
* unable to record the medical data through terminal applications(APP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
adverse clinical events | 2 years
  net adverse clinical events during 2 years follow-up, including death, myocardial infarction, stroke, ischemia induced target vessel revascularization, BARC type 2-5 bleeding
BRAC 2-5 type bleeding | 2 years
  defined as bleeding event graded 2 to 5 of Standardized bleeding definitions from the Bleeding Academic Research Consortium（BRAC）

SECONDARY OUTCOMES:
heart and cerebral vessels ischemia | 2 years
  adeverse events of vascular death, myocardial infarction and stroke
readmission | 2 years
  incidence of readmission during 2-year follow-up
angina recurrence | 2 years
  incidence of angina recurrence during 2-year follow-up
treatment discontinuation | 2 years
  incidence of treatment discontinuation during 2-year follow-up
drug-related events | 2 years
  incidence of drug-related adverse reaction during 2-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, M.D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China